CLINICAL TRIAL: NCT01820689
Title: Tympanometric Analysis in Post Surgical Individuals With Cleft Palate
Brief Title: Tympanometric Analysis in Cleft Palate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Diagnostico Auditivo de Cuiaba (Other)
Collaborators: Federal University of Mato Grosso (Other)
Responsible Party: Principal Investigator, Priscila de Araujo Lucas Rodrigues, Doctor, Centro de Diagnostico Auditivo de Cuiaba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUJM
Record Dates: First submitted 2013-03-18; First posted 2013-03-29 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Bilateral Complete Cleft Lip and/or Alveolus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tympanometry measurement (Experimental)
  Interventions: Other: Tympanometry measurement

INTERVENTIONS:
Other: Tympanometry measurement — The tympanometry measurement will be verify and compared with the time of palatoplasty.

SUMMARY:
Purpose: Characterize the profile of tympanometric patients with cleft lip and palate in the post surgery period and correlate it with the time of palatoplasty. Methods: The sample consisted of 16 patients with cleft lip or palate totaling 32 ears treated at a Public University Hospital in Cuiabá (MT)- Brazil, in the post surgery moment that varied from three months to 33 years. Were sampled patients of both sexes, pediatrics and adults.

ELIGIBILITY:
Inclusion Criteria:

* cleft incisive trans unilateral or bilateral
* post-foramen complete or incomplete

Exclusion Criteria:

* isolated cleft lip
* associated syndromes
* malformation of ear

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Tympanic membrane mobility | 3 months to 33 years
  Tympanic membrane mobility will be measured through the tympanometry and will be demonstrated through their complacency in ml.

SECONDARY OUTCOMES:
Time of palatoplasty | 3 months to 33 years

CONTACTS AND LOCATIONS:
Overall Officials: P A Rodrigues, Doctor, Principal Investigator — HUJM